CLINICAL TRIAL: NCT06649240
Title: Optimal Target Low-density Lipoprotein Cholesterol Level for Small Vessel Occlusion Stroke (SVO70)
Brief Title: Optimal Target Low-density Lipoprotein Cholesterol Level for Small Vessel Occlusion Stroke
Acronym: SVO70
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Hanmi Pharmaceutical co., ltd. (Other)
Responsible Party: Principal Investigator, Seung-Hoon Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-2310-119-1479; KCT0009043 (Registry Identifier: CRIS)
Record Dates: First submitted 2024-10-14; First posted 2024-10-18 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Ischemic Stroke; Small Vessel Cerebrovascular Disease; Cholesterol, LDL; Secondary Prevention; Cardiovascular Diseases
Keywords: Cerebral Small Vessel Diseases; Ischemic Stroke; Secondary Prevention; Cholesterol, LDL; Statins
MeSH Terms: conditions — Ischemic Stroke; Cerebral Small Vessel Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Prospective, Randomized, Open-label, Blinded Endpoint (PROBE) trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive group (Experimental): Target LDL-cholesterol <70 mg/dL
  Interventions: Drug: Statins and/or Ezetimibe; Drug: PCSK9 inhibitor
- Standard group (Active Comparator): Target LDL-cholesterol 90-110 mg/dL
  Interventions: Drug: Statins and/or Ezetimibe; Drug: PCSK9 inhibitor

INTERVENTIONS:
Drug: Statins and/or Ezetimibe — Statin ± Ezetimibe to achieve target LDL-cholesterol level
Drug: PCSK9 inhibitor — The use of PCSK9 inhibitors is permitted to achieve target LDL-cholesterol levels in participants who did not reach the target with statins ± ezetimibe.

SUMMARY:
Lipid-lowering therapy constitutes a cornerstone of secondary prevention in ischemic stroke; however, current stroke guidelines remain deficient in providing optimal target low-density lipoprotein (LDL)-cholesterol levels tailored to the stroke subtypes. Most clinical trials on LDL-cholesterol management have not differentiated between stroke subtypes or have primarily focused on large artery atherosclerosis (LAA) stroke, leaving a gap in evidence for managing LDL-cholesterol in other stroke subtypes, e.g., small vessel occlusion (SVO) stroke. While hypertension is the leading risk factor for SVO strokes, the link between elevated LDL-cholesterol and SVO stroke is also recognized. Establishing optimal LDL-cholesterol targets for SVO stroke would significantly enhance secondary prevention strategies and improve patient outcome. Thus, the investigators aim to compare intensive versus standard lipid-lowering in patients with SVO stroke. SVO70 is a multicenter, prospective, randomized, open, blinded-endpoint clinical trial. Adult participants with objectively confirmed SVO stroke within 180 days of randomization will be included. Exclusion criteria include those with predefined LDL-cholesterol targets for other conditions, statin contraindications, or women who are pregnant, breastfeeding, or planning pregnancy during the study period. Eligible participants will be randomized 1:1 to target LDL-cholesterol <70 mg/dL (intensive group) or 90-110 mg/dL (standard group). The trial plans to enroll 4,016 participants, with the primary outcome being major adverse cardiovascular events-cardiovascular death, stroke, and acute coronary syndrome-during a follow-up period of at least 4 years. This study would provide valuable information for determining the optimal LDL-cholesterol target for patients with SVO stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 years or older
2. Patients with objectively confirmed small vessel occlusive infarctions in the subcortical or brainstem regions, identified through neuroimaging (MRI or CT)
3. Patients with a history of symptomatic ischemic stroke caused by the lesion described in 2), occurring within 180 days prior to enrollment
4. Patients or guardians who agree to the study protocol and sign with informed consent

Exclusion Criteria:

1. Patients requiring intensive LDL cholesterol management (LDL-C <70 mg/dL) due to another condition, with LDL cholesterol targets specified in the guidelines for that condition
2. Patients contraindicated for statin use (e.g., active liver disease, serum transaminase levels elevated more than three times the normal limit, muscle disorders, hypersensitivity to statins, or taking medications contraindicated for use with statins)
3. Women who are pregnant, breastfeeding, or intending to become pregnant during the study period
4. Deemed unsuitable for participation in the study for more than four years, as per the investigators' discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4016 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular event | 4 years
  Major adverse cardiovascular event (MACE) includes cardiovascular death, stroke, and acute coronoary syndrome (i.e., ST-elevation myocardial infarction, non-ST elevation myocardial infarction, and unstable angina).

SECONDARY OUTCOMES:
Any stroke | 4 years
  Ischemic stroke, transient ischemic attack, or hemorrhagic stroke
Ischemic stroke or transient ischemic attack | 4 years
Cardiovascular death | 4 years
Myocardial infarction | 4 years
Any death | 4 years
Acute coronary syndrome | 4 years
  ST-elevation myocardial infarction, non-ST elevation myocardial infarction, and unstable angina

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hoon Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (46):
- South Korea (46):
  - Korea University Ansan Hospital, Ansan
  - Hallym University Sacred Heart Hospital, Anyang
  - Pusan National University Hospital, Busan
  - Gyeongsang National University Changwon Hospital, Changwon
  - Samsung Changwon Hospital, Changwon
  - Chungbuk National University Hospital, Cheongju-si
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon
  - Kangwon National University Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Chilgok Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Daejeon Eulji Medical Center, Daejeon
  - Dongguk University Ilsan Hospital, Goyang
  - Ilsan Paik Hospital, Goyang
  - National Health Insurance Service Ilsan Hospital, Goyang
  - Hanyang University Guri Hospital, Guri-si
  - Chonnam National University Hospital, Gwangju
  - Chosun University Hospital, Gwangju
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong
  - Dongtan Sacred Heart Hospital, Hwaseong
  - Wonkwang University Hospital, Iksan
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - International St. Mary's Hospital, Incheon
  - Jeju National University Hospital, Jeju City
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Hallym University Kangdong Sacred Heart Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Kyung Hee University Medical Center, Seoul
  - National Medical Center, Seoul
  - Nowon Eulji Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Metropolitan Government-Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Yeouido St. Mary's Hospital, Seoul
  - Yongin Severance Hospital, Yŏngin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams HP Jr, Bendixen BH, Kappelle LJ, Biller J, Love BB, Gordon DL, Marsh EE 3rd. Classification of subtype of acute ischemic stroke. Definitions for use in a multicenter clinical trial. TOAST. Trial of Org 10172 in Acute Stroke Treatment. Stroke. 1993 Jan;24(1):35-41. doi: 10.1161/01.str.24.1.35. PMID 7678184
- [Background] Amarenco P, Benavente O, Goldstein LB, Callahan A 3rd, Sillesen H, Hennerici MG, Gilbert S, Rudolph AE, Simunovic L, Zivin JA, Welch KM; Stroke Prevention by Aggressive Reduction in Cholesterol Levels Investigators. Results of the Stroke Prevention by Aggressive Reduction in Cholesterol Levels (SPARCL) trial by stroke subtypes. Stroke. 2009 Apr;40(4):1405-9. doi: 10.1161/STROKEAHA.108.534107. Epub 2009 Feb 19. PMID 19228842
- [Background] Duering M, Biessels GJ, Brodtmann A, Chen C, Cordonnier C, de Leeuw FE, Debette S, Frayne R, Jouvent E, Rost NS, Ter Telgte A, Al-Shahi Salman R, Backes WH, Bae HJ, Brown R, Chabriat H, De Luca A, deCarli C, Dewenter A, Doubal FN, Ewers M, Field TS, Ganesh A, Greenberg S, Helmer KG, Hilal S, Jochems ACC, Jokinen H, Kuijf H, Lam BYK, Lebenberg J, MacIntosh BJ, Maillard P, Mok VCT, Pantoni L, Rudilosso S, Satizabal CL, Schirmer MD, Schmidt R, Smith C, Staals J, Thrippleton MJ, van Veluw SJ, Vemuri P, Wang Y, Werring D, Zedde M, Akinyemi RO, Del Brutto OH, Markus HS, Zhu YC, Smith EE, Dichgans M, Wardlaw JM. Neuroimaging standards for research into small vessel disease-advances since 2013. Lancet Neurol. 2023 Jul;22(7):602-618. doi: 10.1016/S1474-4422(23)00131-X. Epub 2023 May 23. PMID 37236211
- [Background] Goldstein LB, Amarenco P, Szarek M, Callahan A 3rd, Hennerici M, Sillesen H, Zivin JA, Welch KM; SPARCL Investigators. Hemorrhagic stroke in the Stroke Prevention by Aggressive Reduction in Cholesterol Levels study. Neurology. 2008 Jun 10;70(24 Pt 2):2364-70. doi: 10.1212/01.wnl.0000296277.63350.77. Epub 2007 Dec 12. PMID 18077795
- [Background] Mok V, Kim JS. Prevention and Management of Cerebral Small Vessel Disease. J Stroke. 2015 May;17(2):111-22. doi: 10.5853/jos.2015.17.2.111. Epub 2015 May 29. PMID 26060798
- [Background] Hosomi N, Nagai Y, Kohriyama T, Ohtsuki T, Aoki S, Nezu T, Maruyama H, Sunami N, Yokota C, Kitagawa K, Terayama Y, Takagi M, Ibayashi S, Nakamura M, Origasa H, Fukushima M, Mori E, Minematsu K, Uchiyama S, Shinohara Y, Yamaguchi T, Matsumoto M; J-STARS Collaborators. The Japan Statin Treatment Against Recurrent Stroke (J-STARS): A Multicenter, Randomized, Open-label, Parallel-group Study. EBioMedicine. 2015 Aug 6;2(9):1071-8. doi: 10.1016/j.ebiom.2015.08.006. eCollection 2015 Sep. PMID 26501105
- [Background] Amarenco P, Bogousslavsky J, Caplan LR, Donnan GA, Wolf ME, Hennerici MG. The ASCOD phenotyping of ischemic stroke (Updated ASCO Phenotyping). Cerebrovasc Dis. 2013;36(1):1-5. doi: 10.1159/000352050. Epub 2013 Jul 30. PMID 23899749
- [Background] Amarenco P, Kim JS, Labreuche J, Charles H, Abtan J, Bejot Y, Cabrejo L, Cha JK, Ducrocq G, Giroud M, Guidoux C, Hobeanu C, Kim YJ, Lapergue B, Lavallee PC, Lee BC, Lee KB, Leys D, Mahagne MH, Meseguer E, Nighoghossian N, Pico F, Samson Y, Sibon I, Steg PG, Sung SM, Touboul PJ, Touze E, Varenne O, Vicaut E, Yelles N, Bruckert E; Treat Stroke to Target Investigators. A Comparison of Two LDL Cholesterol Targets after Ischemic Stroke. N Engl J Med. 2020 Jan 2;382(1):9. doi: 10.1056/NEJMoa1910355. Epub 2019 Nov 18. PMID 31738483
- [Background] Kleindorfer DO, Towfighi A, Chaturvedi S, Cockroft KM, Gutierrez J, Lombardi-Hill D, Kamel H, Kernan WN, Kittner SJ, Leira EC, Lennon O, Meschia JF, Nguyen TN, Pollak PM, Santangeli P, Sharrief AZ, Smith SC Jr, Turan TN, Williams LS. 2021 Guideline for the Prevention of Stroke in Patients With Stroke and Transient Ischemic Attack: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2021 Jul;52(7):e364-e467. doi: 10.1161/STR.0000000000000375. Epub 2021 May 24. No abstract available. PMID 34024117
- [Background] Amarenco P, Bogousslavsky J, Callahan A 3rd, Goldstein LB, Hennerici M, Rudolph AE, Sillesen H, Simunovic L, Szarek M, Welch KM, Zivin JA; Stroke Prevention by Aggressive Reduction in Cholesterol Levels (SPARCL) Investigators. High-dose atorvastatin after stroke or transient ischemic attack. N Engl J Med. 2006 Aug 10;355(6):549-59. doi: 10.1056/NEJMoa061894. PMID 16899775
- [Background] Kim JY, Kang K, Kang J, Koo J, Kim DH, Kim BJ, Kim WJ, Kim EG, Kim JG, Kim JM, Kim JT, Kim C, Nah HW, Park KY, Park MS, Park JM, Park JH, Park TH, Park HK, Seo WK, Seo JH, Song TJ, Ahn SH, Oh MS, Oh HG, Yu S, Lee KJ, Lee KB, Lee K, Lee SH, Lee SJ, Jang MU, Chung JW, Cho YJ, Choi KH, Choi JC, Hong KS, Hwang YH, Kim SE, Lee JS, Choi J, Kim MS, Kim YJ, Seok J, Jang S, Han S, Han HW, Hong JH, Yun H, Lee J, Bae HJ. Executive Summary of Stroke Statistics in Korea 2018: A Report from the Epidemiology Research Council of the Korean Stroke Society. J Stroke. 2019 Jan;21(1):42-59. doi: 10.5853/jos.2018.03125. Epub 2018 Dec 18. PMID 30558400